CLINICAL TRIAL: NCT04524286
Title: The Role of a Midwifery Continuity of CARE Model in Reducing Health Inequalities in Childbearing Women and Babies Living on a Low-income: The Mi-CARE Study
Brief Title: Role of Midwifery Continuity of Care in Reducing Health Inequalities
Acronym: Mi-CARE
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19/20/IRAS/CC; 262369 (Other: IRAS); 45534 (Other: CPMS)
Record Dates: First submitted 2020-08-14; First posted 2020-08-24 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Health Knowledge, Attitudes, Practice; Social Determinants; Public Health; Pregnancy Related
Keywords: Midwifery Continuity of Care; Social Determinants of Health; Childbearing women; Health inequalities/inequities; Constructivist Grounded Theory; Qualitative research
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Public - Childbearing Women: Childbearing women living in three deprived areas in a city in the South of England.
  Interventions: Other: Interviews only.
- Staff - Midwives: Midwives working in caseloading teams providing continuity of care to women living in three deprived areas in a city in the South of England.
  Interventions: Other: Interviews only.

INTERVENTIONS:
Other: Interviews only. — Interviews will be conducted with childbearing women and midwives.

SUMMARY:
The impact of living in a deprived area has far reaching consequences on maternal and infant health. Studies in England show women living in deprived areas have some of the poorest experiences of care, poor birth outcomes and are 50% more likely to die of pregnancy related complications than women in the least deprived neighbourhoods. Life expectancy has also stalled for women living in the most deprived areas and the global COVID-19 pandemic has further amplified existing health inequalities.

The Social Determinants of Health (SDH) are the conditions in which people are born, grow, work, live, and age, and are mostly responsible for health inequities - the unfair and avoidable differences in health seen within and between populations. Evidence shows taking action on the SDH alongside Midwifery Continuity of Care (MCC) models, improves birth outcomes and reduces health inequalities. How midwives working in MCC models in areas of high deprivation address the SDH as part of their public health and prevention role is currently not clear. There is also a lack of qualitative evidence exploring the SDH from the perspectives of women themselves.

Drawing on Constructivist Grounded Theory methods, this research will take place in a low-income setting in England. Through the use of semi-structured interviews with women and midwives working in an NHS MCC model, the study will generate theory to help explain how and indeed whether midwives take action to address the SDH as part of their public health role. The study also seeks to understand the SDH impacting upon women's lives and what mechanisms exist to support or obstruct engagement with the SDH. Examining these domains will contribute to the evidence base about the impact of MCC and the public health and prevention strategy in NHS maternity services.

ELIGIBILITY:
Inclusion Criteria - Childbearing Women

* Women who are currently receiving maternity care from the MCC caseloading teams;
* Women who have previously received care from one of the caseloading teams;
* Women aged 16 and over;
* Women who can understand English and are able to independently provide their informed consent;
* Women at any point in their pregnancy or up to five years following the birth of their babies. This time frame is considered appropriate in order to capture women who are currently receiving maternity care and those who have received care locally in the last five years. This will aim to also capture women's experiences before referral to the caseloading teams changed;
* Women who had or are currently having their maternity care provided by UHS.

Inclusion Criteria - Midwives

* Midwives who work in the MCC caseloading teams in the study setting;
* Midwives who have previously worked in the local MCC caseloading teams.
* Midwifery managers who have managerial oversight of the MCC caseloading teams.

Exclusion Criteria - Childbearing women

* Women who have not received care from one of the MCC caseloading teams;
* Women who gave birth more than five years ago;
* Women below the age of 16 years;
* Women who cannot speak English due to a lack of financial resources to fund translation services;
* Women who are in labour;
* Women who had their maternity care at a different NHS Trust;
* Women who lack capacity to provide informed consent;
* Women who decline to participate and decline to provide informed consent.

Exclusion criteria - Midwives

* Midwives who work in the universal teams;
* MSWs due to different professional roles and responsibilities;
* Midwives who decline to participate and decline to provide informed consent.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * Childbearing women - Women who receive their care from one of the MCC caseloading teams. In the context of this study the term 'childbearing woman' is defined as any woman of childbearing age over the age of 16 years who is currently pregnant or up to five years post childbirth;
  * Midwives - Midwives working in the study setting or have worked in one of the MCC caseloading teams. Also, midwives at the study site who have managerial and leadership oversight of the MCC teams.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Interviews with childbearing women | 12 months
  Women living in the case setting willing to participate and share their maternity care experiences in one-to-one interviews.
Interviews with childbearing women | 12 months
  Women living in the case setting willing to participate and share their childbearing experiences in one-to-one interviews.
Interview with midwives | 12 months
  Midwives willing to participate and share their experiences of providing care to women in the case setting.
Interview with midwives | 12 months
  Midwives willing to participate and share their knowledge about their public health role and how the actions they take to meet the needs of women.

SECONDARY OUTCOMES:
Document analysis | 12 months
  Analysis of documents such as policies, reports and guidelines which focus on maternal health inequalities, the public health role of midwives, and the role of midwifery-led continuity of care.
Memo writing | 12 months
  Memos will be written throughout data collection and incorporated into data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Clayton, Principal Investigator — Bournemouth University
Locations (1):
- Princess Anne Hospital - University Hospital Southampton, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will be anonymised, cleaned and stored within Bournemouth University's online research data repository BORDaR. This is a central location where research data generated by Bournemouth University is stored. This is accessible to the public for reuse.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: After the study has ended and for 25 years after this.
URL: http://bordar.bournemouth.ac.uk/